CLINICAL TRIAL: NCT05529472
Title: KAIZEN: Safety and Effectiveness Evaluation of Peripheral Orbital Atherectomy
Brief Title: Safety and Effectiveness Evaluation of Peripheral Orbital Atherectomy
Acronym: KAIZEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-0013-P
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Artery Disease
Keywords: superficial femoral artery; popliteal artery; de novo lesions
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Peripheral Orbital Atherectomy System (OAS) (Experimental): Treatment with Cardiovascular Systems, Inc. (CSI) Orbital Atherectomy System (OAS) followed by Percutaneous Old Balloon Angioplasty (POBA) pre-dilation and Medtronic IN.PACT™ Admiral™ Drug Coated Balloon (DCB)
  Interventions: Device: Peripheral Orbital Atherectomy System (OAS)

INTERVENTIONS:
Device: Peripheral Orbital Atherectomy System (OAS) — Treatment with Orbital Atherectomy System (OAS) followed by Percutaneous Old Balloon Angioplasty (POBA), pre-dilation and Drug Coated Balloon (DCB) - Medtronic IN.PACT™ Admiral™

SUMMARY:
This is a prospective, single-arm, multi-center study designed to evaluate the safety and efficacy of the Orbital Atherectomy System (OAS) for the treatment of adult Japanese subjects with a de novo symptomatic calcified occlusive atherosclerotic lesion in the superficial femoral artery (SFA) and/or popliteal (POP) artery, which would be otherwise ineligible for endovascular therapy due to risk of complication. Study objective is to collect safety and effectiveness data to support potential commercialization of the peripheral OAS device in Japan.

ELIGIBILITY:
General Inclusion Criteria (≤30 Days from Clinical Trial Treatment):

* 18 years of age or older
* Subject has signed the approved KAIZEN study Informed Consent Form prior to any study-related procedures
* Chronic, symptomatic lower limb ischemia
* Clinical indication for percutaneous transluminal angioplasty intervention in the native SFA and/or POP artery

General Exclusion Criteria (≤30 Days from Clinical Trial Treatment):

* Female who is pregnant and/or breastfeeding
* Currently participating in another investigational clinical study
* Unwilling to follow the Investigator's instructions or follow-up requirements
* Any non-diagnostic peripheral vascular intervention that was unsuccessful or had complications within 30 days before clinical trial treatment
* Any non-diagnostic coronary intervention within 30 days before clinical trial treatment
* Any planned non-diagnostic vascular intervention(s) within 30 days after clinical trial treatment
* Any planned procedures or other medical conditions which, in the Investigator's opinion, may interfere with the study result and/or subject's optimal participation in the study
* Prior major amputation within one year of the clinical trial treatment procedure
* Planned major amputation
* Life expectancy of ≤6 months
* History of coagulopathy or hypercoagulable bleeding disorder
* History of Myocardial Infarction (MI), or stroke/cerebrovascular accident within 6-months prior to the clinical trial treatment
* Unstable angina pectoris
* Untreatable hemorrhagic disease or platelet count <80,000mm3 or >600,000mm3
* Evidence of active infection
* Known hypersensitivity or contraindication to contrast dye
* Known hypersensitivity/allergy to the investigational atherectomy system or protocol-related therapies
* Known contraindication to antiplatelet therapy
* Creatinine > 2.5 mg/dL, unless on dialysis

Clinical Trial Treatment Inclusion:

* De novo target lesion
* All guidewires cross the target lesion within the true lumen
* Target lesion with ≥70% stenosis
* Target reference vessel diameter (RVD) ≥3.0 mm and ≤6.0 mm
* Target lesion length ≤150 mm
* Minimum one patent tibial vessel on the target leg
* Target lesion has visual evidence of calcification

Clinical Trial Treatment Exclusion:

* Any inflow treatment that was unsuccessful or had complications during the clinical trial treatment, prior to subject enrollment
* Target lesion is a chronic total occlusion
* Presence of any other lesions in the target limb requiring a planned surgical intervention or endovascular procedure 30-days after clinical trial treatment
* Presence of aneurysm in the target vessel
* Acute ischemia and/or acute thrombosis of the SFA and/or POP artery
* Angiographic evidence of perforation
* Angiographic evidence of severe dissection
* Planned use of atherectomy other than Cardiovascular Systems, Inc. (CSI) Peripheral OAS in the target limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroyoshi Yokoi, MD, Principal Investigator — International University of Health and Welfare, Japan
Locations (12):
- Japan (12):
  - Tokyo bay Ichikawa, Urayasu, Chiba
  - Matsuyama Red Cross, Matsuyama, Ehime
  - Fukuoka Sannou, Sawara, Fukuoka
  - Iwaki-City Medical Center, Iwaki, Fukushima
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Kyoto Katsura Hospital, Nishikyo-ku, Kyoto
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Nara Medical University, Kashihara, Nara
  - Morinomiya, Joto, Osaka
  - Ageo Central Hospital, Ageo, Saitama
  - Kasukabe Central (Chu-o-), Kasukabe, Saitama
  - Daini Osaka Police Hospital, Osaka

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 81 subjects were enrolled at 12 Japanese sites between 10January2023 and 19March2024 with 14 subjects in roll-in cohort and 67 in full analysis set (FAS). Subjects were considered to enrolled in study at time point of Peripheral Orbital Atherectomy System (OAS) guide wire entered body and became part of ITT population (N=67). 66 subjects became mITT population,1could not confirm calcification due to insufficient imaging. All 14 roll-in subjects were analyzed separately from enrolled population.
Pre-assignment Details: The 14 subjects enrolled in a roll-in cohort, were conducted as part of the site initiation phase to allow operating investigators for procedural training with the investigational device. These roll-in subjects were not included in the Full Analysis Set (FAS) and were not part of the reported results in Participant Flow, Baseline Characteristics, Outcome Measures, or Adverse Events modules, as predefined in the statistical analysis plan.
Groups:
- Analysis Cohort [Peripheral Orbital Atherectomy System (OAS)]: Treatment with Cardiovascular Systems, Inc. (CSI) Orbital Atherectomy System (OAS) followed by Percutaneous Old Balloon Angioplasty (POBA) pre-dilation and Medtronic IN.PACT™ Admiral™ Drug Coated Balloon (DCB)
  Peripheral Orbital Atherectomy System (OAS): Treatment with Orbital Atherectomy System (OAS) followed by Percutaneous Old Balloon Angioplasty (POBA), pre-dilation and Drug Coated Balloon (DCB) - Medtronic IN.PACT™ Admiral™
- Roll-in Cohort [Peripheral Orbital Atherectomy System(OAS)]: Roll-in subjects were initial cases by the investigator enrolled to ensure proper device training, and procedural and data collection adherence. Roll-in subjects were consented, treated, and followed per protocol. Roll-in subject data was reported and analyzed separately from the Analysis Cohort.
Period: Overall Study
Arm/Group | Analysis Cohort [Peripheral Orbital Atherectomy System (OAS)] | Roll-in Cohort [Peripheral Orbital Atherectomy System(OAS)]
Started | 67 | 14
Completed | 66 | 13
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Analysis Cohort[Peripheral Orbital Atherectomy System(OAS)]: Treatment with Cardiovascular Systems, Inc. (CSI) Orbital Atherectomy System (OAS) followed by Percutaneous Old Balloon Angioplasty (POBA) pre-dilation and Medtronic IN.PACT™ Admiral™ Drug Coated Balloon (DCB)
  Peripheral Orbital Atherectomy System (OAS): Treatment with Orbital Atherectomy System (OAS) followed by Percutaneous Old Balloon Angioplasty (POBA), pre-dilation and Drug Coated Balloon (DCB) - Medtronic IN.PACT™ Admiral™
- Total: Total of all reporting groups
Arm/Group | Analysis Cohort[Peripheral Orbital Atherectomy System(OAS)] | Roll-in Cohort [Peripheral Orbital Atherectomy System(OAS)] | Total
Number analyzed (Participants) | 67 | 14 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.6 (7.51) | 73.6 (7.91) | 74.6 (7.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 3 | 23
  Male | 47 | 11 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 67 | 14 | 81
Body mass index [Mean (Standard Deviation); unit: kg/m²] | 23.1 (3.61) | 24.2 (3.68) | 23.65 (3.64)
Rutherford classification [Count of Participants; unit: Participants] — Rutherford Classification: Class 0 : Asymptomatic; no hemodynamically significant occlusive disease. Class 1: Mild Claudication; there is no limitation with ordinary physical activities. Class 2: Moderate Claudication; there is a slight limitation of ordinary physical activities. Class 3: Severe Claudication; there is marked limitation of ordinary physical activities. Class 4: Ischemic rest pain. Class5:Minor tissue loss, non-healing ulcer, focal gangrene with diffuse pedal ischemia. Class6: Major tissue loss extending above transmetatarsal level; functional foot no longer salvageable.
  Participants
    Moderate Claudication (RC2) | 20 | 6 | 26
    Severe Claudication (RC3) | 39 | 8 | 47
    Ischemic rest pain (RC4) | 8 | 0 | 8
Serum Creatinine [Mean (Standard Deviation); unit: mg/dl] | 3.1 (3.12) | 3.5 (3.79) | 3.3 (3.45)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Acute Device Success
Description: The percentage of subjects with the following, post-procedure:
  1. ≤50% residual stenosis post OAD + POBA [Angiographic Core Lab assessed] and,
  2. No OAS-related severe angiographic complications defined as severe dissections (D-F), perforation, or distal emboli requiring additional treatment during the procedure [CEC adjudicated].
Time Frame: At the end of the procedure
Population: The mITT population set included all enrolled subjects who have been treated with the OAD on a target lesion that has met Independent Physician Review, regardless of deviations from the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Analysis Cohort[Peripheral Orbital Atherectomy System(OAS)]
Number analyzed (Participants) | 66
Participants | 55

2. Secondary Outcome: Change in Lesion Stenosis
Description: The percentage changes in diameter stenosis of the target lesion at each stage of the procedure: Baseline, Post OAD, Post POBA and Post DCB [Angiographic Core Lab assessed].
Time Frame: Baseline, Post OAD, Post POBA
Population: The ITT population included all enrolled 67 subjects who have been treated with the OAD regardless of deviations from the protocol. The mITT population set included all enrolled subjects who have been treated with the OAD on a target lesion that has met Independent Physician Review, regardless of deviations from the protocol. Of 67 enrolled subjects, one could not confirm calcification due to insufficient imaging, resulting in mITT analysis population becoming 66 subjects
Measure: Mean (Standard Deviation); unit: percentage of stenosis
Arm/Group | Analysis Cohort[Peripheral Orbital Atherectomy System(OAS)]
Number analyzed (Participants) | 67
percentage of stenosis
  Baseline (ITT population) | 73.7 (14.54)
  Post final OAD (ITT population): number analyzed (Participants) | 65
  Post final OAD (ITT population) | 47.8 (11.96)
  Post POBA (ITT population) | 23.2 (10.25)
  Reduction in % Diameter Stenosis (Pre-procedure - Post OAD) (ITT population): number analyzed (Participants) | 65
  Reduction in % Diameter Stenosis (Pre-procedure - Post OAD) (ITT population) | 25.9 (14.89)
  Reduction in % Diameter Stenosis (Pre-procedure - Post POBA) (ITT population) | 50.5 (17.80)
  Baseline (mITT population): number analyzed (Participants) | 66
  Baseline (mITT population) | 73.7 (14.65)
  Post final OAD (mITT population): number analyzed (Participants) | 66
  Post final OAD (mITT population) | 47.9 (12.04)
  Post POBA (mITT population): number analyzed (Participants) | 66
  Post POBA (mITT population) | 23.1 (10.31)
  Reduction in % Diameter Stenosis (Pre-procedure - Post OAD) (mITT population): number analyzed (Participants) | 66
  Reduction in % Diameter Stenosis (Pre-procedure - Post OAD) (mITT population) | 25.8 (14.99)
  Reduction in % Diameter Stenosis (Pre-procedure - Post POBA) (mITT population): number analyzed (Participants) | 66
  Reduction in % Diameter Stenosis (Pre-procedure - Post POBA) (mITT population) | 50.5 (17.93)

3. Secondary Outcome: Acute Technical Success
Description: Acute technical success defined per the Peripheral Academic Research Consortium (PARC) definition of achievement of a final residual stenosis <30% for stented and <50% for non-stented subjects by angiography at the end of the procedure [Angiographic Core Lab assessed] without severe angiographic complications defined as severe dissections (D-F), perforation, or distal emboli requiring additional treatment during the procedure [CEC adjudicated].
Time Frame: At the end of the procedure
Population: The ITT population included all enrolled 67 subjects who have been treated with the OAD regardless of deviations from the protocol. The mITT population set included all enrolled subjects who have been treated with the OAD on a target lesion that has met Independent Physician Review, regardless of deviations from the protocol. Of enrolled 67 subjects, one could not confirm calcification due to insufficient imaging, resulting in mITT analysis population becoming 66 subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Analysis Cohort[Peripheral Orbital Atherectomy System(OAS)]
Number analyzed (Participants) | 67
Participants
  ITT population | 56
  mITT population: number analyzed (Participants) | 66
  mITT population | 55

4. Secondary Outcome: Drug Coated Balloon (DCB) Device Success
Description: DCB Device Success defined as the ability to achieve successful delivery and deployment of all DCB to the target lesion as described per the Instructions for Use (IFU) within 3 minutes of insertion without removal and use of an additional device.
Time Frame: Within 3 minutes of insertion of DCB
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Analysis Cohort[Peripheral Orbital Atherectomy System(OAS)]
Number analyzed (Participants) | 67
percentage of participants
  ITT Population | 98.5 [92.0 to 100.0]
  mITT population: number analyzed (Participants) | 66
  mITT population | 98.5 [91.8 to 100.0]

5. Secondary Outcome: Target Vessel Patency
Description: Target Vessel Patency is a binary composite endpoint comprised of:
  * CEC adjudicated absence of clinically driven repeat procedure performed for ≥50% stenosis confirmed by angiography within all or part of the target lesion after documentation of recurrent clinical symptoms of PAD following clinical trial treatment procedure (i.e. clinically-driven TLR) occurring at any time-point on, or prior to the 6-month visit date and,
  * a Duplex Ultrasound Core Lab assessed PSVR value of ≤2.4 (or equivalent by visual assessment if the lesion is non-patent and the PSVR cannot be numerically calculated).
  The vessel is considered patent if both criteria are met at the time of assessment.
Time Frame: Up to 6 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Analysis Cohort[Peripheral Orbital Atherectomy System(OAS)]
Number analyzed (Participants) | 67
percentage of participants
  ITT population | 92.3 [83.0 to 97.5]
  mITT population: number analyzed (Participants) | 66
  mITT population | 92.2 [82.7 to 97.4]

6. Secondary Outcome: Rate of Severe Angiographic Complications
Description: Rate of severe angiographic complications defined as severe dissections (D-F), perforation, or distal emboli requiring additional treatment during the procedure [CEC adjudicated]
Time Frame: At the end of the procedure
Population: The FAS population included all subjects enrolled into the trial regardless of treatment with the OAD or deviations from the protocol. The mITT population set included all enrolled subjects who have been treated with the OAD on a target lesion that has met Independent Physician Review, regardless of deviations from the protocol. Of 67 enrolled subjects, one could not confirm calcification due to insufficient imaging, resulting in mITT analysis population becoming 66 subjects
Measure: Number; unit: participants
Arm/Group | Analysis Cohort[Peripheral Orbital Atherectomy System(OAS)]
Number analyzed (Participants) | 67
participants
  Dissection (D-F): FAS population | 0
  Perforation: FAS population | 1
  Distal Emboli: FAS population | 10
  Dissection (D-F): mITT population: number analyzed (Participants) | 66
  Dissection (D-F): mITT population | 0
  Perforation: mITT population: number analyzed (Participants) | 66
  Perforation: mITT population | 1
  Distal Emboli: mITT population: number analyzed (Participants) | 66
  Distal Emboli: mITT population | 10

7. Secondary Outcome: Acute Procedural Success
Description: Acute procedural success is defined as both acute technical success and absence of death, stroke, myocardial infarction (MI), acute onset of limb ischemia, index bypass graft or treated segment thrombosis, and/or need for urgent/emergent vascular surgery within 72 hours of the clinical trial treatment [CEC adjudicated].
Time Frame: 72 hours after index procedure
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Analysis Cohort[Peripheral Orbital Atherectomy System(OAS)]
Number analyzed (Participants) | 67
percentage of participants
  FAS population | 83.6 [72.5 to 91.5]
  mITT population: number analyzed (Participants) | 66
  mITT population | 83.3 [72.1 to 91.4]

8. Secondary Outcome: Rate of Major Adverse Event (MAE)
Description: Major Adverse Event (MAE) rate at 30 days and 6 months (CEC adjudicated) was defined as:
  1. All-cause death through 30 days or
  2. Major amputation of the target limb or
  3. Clinically-driven TLR
Time Frame: 30 days and 6 months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Analysis Cohort[Peripheral Orbital Atherectomy System(OAS)]
Number analyzed (Participants) | 67
Participants
  30 days (FAS population) : All-cause death | 0
  30 days (FAS population) : Major amputation of the target limb | 0
  30 days (FAS population) : Clinically driven TLR | 0
  6 months (FAS population) : All-cause death | 0
  6 months (FAS population) : Major amputation of the target limb | 0
  6 months (FAS population) : Clinically driven TLR | 1
  30 days (mITT population) : All-cause death: number analyzed (Participants) | 66
  30 days (mITT population) : All-cause death | 0
  30 days (mITT population) : Major amputation of the target limb: number analyzed (Participants) | 66
  30 days (mITT population) : Major amputation of the target limb | 0
  30 days (mITT population) : Clinically driven TLR: number analyzed (Participants) | 66
  30 days (mITT population) : Clinically driven TLR | 0
  6 months (mITT population) : All-cause death: number analyzed (Participants) | 66
  6 months (mITT population) : All-cause death | 0
  6 months (mITT population) : Major amputation of the target limb: number analyzed (Participants) | 66
  6 months (mITT population) : Major amputation of the target limb | 0
  6 months (mITT population) : Clinically driven TLR: number analyzed (Participants) | 66
  6 months (mITT population) : Clinically driven TLR | 1

9. Secondary Outcome: Change of Rutherford Classification (ITT Population)
Description: Rutherford Classification; Class 0: Asymptomatic; no hemodynamically significant occlusive disease.
  Class 1: Mild Claudication; there is no limitation with ordinary physical activities (e.g., walking several blocks, climbing stairs). Limiting symptoms may occur with marked exertion (e.g., strenuous, rapid or prolonged exertion at work or recreation).
  Class 2: Moderate Claudication; there is a slight limitation of ordinary physical activities (e.g., walking uphill, or more than two level blocks, or climbing stairs rapidly). Subject is comfortable at rest.
  Class 3: Severe Claudication; there is marked limitation of ordinary physical activities (e.g., walking 1-2 level blocks or climbing one flight of stairs). Subject is comfortable at rest.
  Class 4: Ischemic rest pain. Class 5: Minor tissue loss, non-healing ulcer, focal gangrene with diffuse pedal ischemia.
  Class 6: Major tissue loss extending above transmetatarsal level; functional foot no longer salvageable.
Time Frame: Baseline, 30 days and 6 months
Population: Analysis population includes all enrolled ITT (intent to treat) subjects who have been treated with the OAD regardless of deviations from the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Analysis Cohort[Peripheral Orbital Atherectomy System(OAS)]
Number analyzed (Participants) | 67
Participants
  Baseline: Grade 0: Asymptomatic (0) | 0
  Baseline: Grade II :Ischemic Rest Pain (4) | 8
  Baseline: Grade III :Minor Tissue Loss (5) | 0
  Baseline: Grade I:Severe Claudication (3) | 39
  Baseline: Grade I:Moderate Claudication (2) | 20
  Baseline: Grade I:Mild Claudication (1) | 0
  30 Days: number analyzed (Participants) | 61
  30 Days: Grade 0: Asymptomatic (0) | 52
  30 Days: Grade I:Moderate Claudication (2) | 1
  30 Days: Grade II :Ischemic Rest Pain (4) | 0
  30 Days: Grade III :Minor Tissue Loss (5) | 0
  30 Days: Grade I:Mild Claudication (1) | 7
  30 Days: Grade I:Severe Claudication (3) | 1
  6 Months: number analyzed (Participants) | 65
  6 Months: Grade 0: Asymptomatic (0) | 55
  6 Months: Grade I:Severe Claudication (3) | 0
  6 Months: Grade I:Mild Claudication (1) | 7
  6 Months: Grade II :Ischemic Rest Pain (4) | 0
  6 Months: Grade III :Minor Tissue Loss (5) | 2
  6 Months: Grade I:Moderate Claudication (2) | 1

10. Secondary Outcome: Change of Rutherford Classification (mITT Population)
Description: as for outcome 9
Time Frame: Baseline, 30 days and 6 months
Population: The mITT analysis set included all enrolled subjects who have been treated with the OAD on a target lesion that has met Independent Physician Review, regardless of deviations from the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Analysis Cohort[Peripheral Orbital Atherectomy System(OAS)]
Number analyzed (Participants) | 66
Participants
  Baseline: Grade 0: Asymptomatic (0) | 0
  Baseline: Grade II :Ischemic Rest Pain (4) | 8
  Baseline: Grade I:Moderate Claudication (2) | 19
  Baseline: Grade III :Minor Tissue Loss (5) | 0
  Baseline: Grade I:Mild Claudication (1) | 0
  Baseline: Grade I:Severe Claudication (3) | 39
  30 Days: number analyzed (Participants) | 60
  30 Days: Grade 0: Asymptomatic (0) | 51
  30 Days: Grade I:Mild Claudication (1) | 7
  30 Days: Grade III :Minor Tissue Loss (5) | 0
  30 Days: Grade II :Ischemic Rest Pain (4) | 0
  30 Days: Grade I:Severe Claudication (3) | 1
  30 Days: Grade I:Moderate Claudication (2) | 1
  6 Months: number analyzed (Participants) | 64
  6 Months: Grade 0: Asymptomatic (0) | 54
  6 Months: Grade II :Ischemic Rest Pain (4) | 0
  6 Months: Grade I:Moderate Claudication (2) | 1
  6 Months: Grade III :Minor Tissue Loss (5) | 2
  6 Months: Grade I:Severe Claudication (3) | 0
  6 Months: Grade I:Mild Claudication (1) | 7

11. Secondary Outcome: Change in Ankle Brachial Index (ABI)
Description: The Ankle-Brachial Index (ABI) is a simple, non-invasive test used to assess peripheral artery disease (PAD). It compares the blood pressure measured at the ankle with the blood pressure measured at the arm (brachial artery).
Time Frame: Baseline (within 30 days of the clinical treatment), and Post Procedure (after the clinical trial treatment prior to discharge: post procedure ABI was collected on average 1.1 days post clinical trial treatment)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Analysis Cohort[Peripheral Orbital Atherectomy System(OAS)]
Number analyzed (Participants) | 67
ratio
  Baseline mean ABI (ITT population): number analyzed (Participants) | 65
  Baseline mean ABI (ITT population) | 0.76 (0.214)
  Post Procedure mean ABI (ITT population): number analyzed (Participants) | 65
  Post Procedure mean ABI (ITT population) | 0.91 (0.178)
  Change in mean ABI (post-procedure - baseline)(ITT population): number analyzed (Participants) | 63
  Change in mean ABI (post-procedure - baseline)(ITT population) | 0.15 (0.186)
  Baseline mean ABI (mITT population): number analyzed (Participants) | 64
  Baseline mean ABI (mITT population) | 0.76 (0.213)
  Post Procedure mean ABI (mITT population): number analyzed (Participants) | 64
  Post Procedure mean ABI (mITT population) | 0.91 (0.179)
  Change in mean ABI (post-procedure - baseline)(mITT population): number analyzed (Participants) | 62
  Change in mean ABI (post-procedure - baseline)(mITT population) | 0.15 (0.187)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Analysis Cohort[Peripheral Orbital Atherectomy System(OAS)] | Roll-in Cohort [Peripheral Orbital Atherectomy System(OAS)]
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/14
Serious Adverse Events (participants affected / at risk) | 27/67 | 5/14
Other Adverse Events (participants affected / at risk) | 49/67 | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Analysis Cohort[Peripheral Orbital Atherectomy System(OAS)] (N=67) | Roll-in Cohort [Peripheral Orbital Atherectomy System(OAS)] (N=14)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cancer (General disorders) | 1 (1) | 1 (1)
Cardiac dysfunction - Chronic heart failure or aggravated (Cardiac disorders) | 1 (1) | 0 (0)
New/worsening claudication (Infections and infestations) | 1 (1) | 0 (0)
New/worsening gangrene (Infections and infestations) | 2 (2) | 0 (0)
New/worsening ulcer (Infections and infestations) | 3 (3) | 0 (0)
Peripheral artery abrupt closure (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery pseudoaneurysm (Vascular disorders) | 1 (1) | 2 (2)
Peripheral artery restenosis (Vascular disorders) | 1 (2) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 3 (3) | 0 (0)
Peripheral artery vasospasm (Vascular disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Spinal cord/nerve root disorders (Nervous system disorders) | 1 (1) | 0 (0)
Other vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Other infection- Localized (Infections and infestations) | 1 (1) | 1 (1)
Adverse event - Other (General disorders) | 3 (3) | 0 (0)
Perforation (Vascular disorders) | 1 (1) | 1 (1)
Distal Emboli (Vascular disorders) | 9 (9) | 0 (0)
Acute onset limb ischemia (Vascular disorders) | 1 (1) | 0 (0)
Dissection (Vascular disorders) | 0 (0) | 1 (1)
Bleeding/hemorrhage, non access site (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Analysis Cohort[Peripheral Orbital Atherectomy System(OAS)] (N=67) | Roll-in Cohort [Peripheral Orbital Atherectomy System(OAS)] (N=14)
Peripheral artery slow flow (Vascular disorders) | 2 (2) | 0 (0)
Peripheral artery vasospasm (Vascular disorders) | 2 (2) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery abrupt closure (Vascular disorders) | 2 (2) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Dissection (Vascular disorders) | 41 (41) | 9 (10)
Perforation (Vascular disorders) | 1 (1) | 1 (1)
Distal Emboli (Vascular disorders) | 16 (16) | 2 (2)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Nausea/vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peripheral arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Site/investigator shall not divulge data or any other information disclosed by Sponsor or CRO in connection with this clinical study or information obtained as a result of this clinical trial to a third party without the prior written consent of Sponsor.
* Site/investigator shall obtain the prior written consent of Sponsor before presenting any information obtained from this clinical trial to the professional academic society or other outside organization.

DOCUMENTS (2):
  • Study Protocol (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT05529472/Prot_002.pdf
  • Statistical Analysis Plan (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/72/NCT05529472/SAP_003.pdf